CLINICAL TRIAL: NCT04969900
Title: Effects of Aromatherapy on Patient Satisfaction With Surgical Abortion at Less Than 10 Weeks Gestation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 21-2561
Record Dates: First submitted 2021-06-25; First posted 2021-07-21 (Actual); Results first posted 2025-08-03 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Surgical Abortion; Patient Satisfaction; Anesthesia; Pain
MeSH Terms: conditions — Patient Satisfaction; Pain | interventions — lavender oil

STUDY DESIGN:
Intervention Model Description: A single-site, double-blinded, placebo-controlled clinical trial of lavender aromatherapy versus inert oil placebo for patient satisfaction in adult women having a first trimester outpatient surgical abortion before 10 weeks and 0 days gestation.
Who Masked: Participant, Care Provider, Investigator
Masking Description: For purposes of masking, all patients enrolled in the study will be required to wear a cloth face covering over their nose and mouth during their procedure to minimize diffusion of the aromatic scent in the procedure room.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo - Jojoba Oil (100% organic golden expeller-pressed Simmondsia chinensis) (Placebo Comparator): Study randomization to lavender aromatherapy or placebo will occur just prior to the initiation of the abortion procedure. A permutated block stratified randomization scheme will be utilized so that equal numbers of participants receiving no sedation and PO sedation will be randomized to lavender aromatherapy or placebo. 1cc of dilute lavender aromatherapy and placebo will be pre-filled in a 5/8 dram mini amber glass bottle provided to the patient. Immediately prior to procedure start (defined as after receiving antibiotic and emptying bladder), participants will be instructed to self-administer the study product. They will bring down their personal cloth mask to chin level and rub the study product within the amber glass bottle on their upper lip and nose (left and right ala, alarfacial grooves, and columella). Participants will be instructed to take 4 deep breaths and then replace their mask over their nose. The patient will then proceed to the procedure.
  Interventions: Other: Placebo oil
- Investigational Product - A 10% dilute Lavandula angustifolia - jojoba oil essential oil blend (Active Comparator): Study randomization to lavender aromatherapy or placebo will occur just prior to the initiation of the abortion procedure. A permutated block stratified randomization scheme will be utilized so that equal numbers of participants receiving no sedation and PO sedation will be randomized to lavender aromatherapy or placebo. 1cc of dilute lavender aromatherapy and placebo will be pre-filled in a 5/8 dram mini amber glass bottle provided to the patient. Immediately prior to procedure start (defined as after receiving antibiotic and emptying bladder), participants will be instructed to self-administer the study product. They will bring down their personal cloth mask to chin level and rub the study product within the amber glass bottle on their upper lip and nose (left and right ala, alarfacial grooves, and columella). Participants will be instructed to take 4 deep breaths and then replace their mask over their nose. The patient will then proceed to the procedure.
  Interventions: Other: Lavender oil.

INTERVENTIONS:
Other: Placebo oil — The placebo group will receive placebo oil.
  Arms: Placebo - Jojoba Oil (100% organic golden expeller-pressed Simmondsia chinensis)
Other: Lavender oil. — Investigational Product. This group will receive Lavender oil.
  Arms: Investigational Product - A 10% dilute Lavandula angustifolia - jojoba oil essential oil blend

SUMMARY:
The investigators propose a single-site, double-blinded, placebo-controlled clinical trial of lavender aromatherapy versus placebo for patient satisfaction in adult women having a surgical abortion before 10 weeks and 0 days gestation. The investigators will evaluate whether lavender aromatherapy is an effective adjunct therapy for patient satisfaction during first trimester surgical abortion. The investigators will measure satisfaction using the Iowa Satisfaction with Anesthesia Scale (ISAS). The investigators hypothesize that women receiving lavender aromatherapy will report higher satisfaction scores compared to women receiving placebo.

Prior studies have investigated the use of aromatherapy in laboring patients, in menstruating women, and in general post-operative populations. No investigations have focused on the use of lavender aromatherapy as an adjunct therapy to paracervical block and/or oral narcotics and anxiolytics in outpatient surgical abortion. Our study is novel in investigating patient satisfaction with first trimester surgical abortion using lavender aromatherapy.

The contribution of this proposed research to the literature is significant because current affordable anesthetic adjuncts to opioids and benzodiazepines are limited.

DETAILED DESCRIPTION:
The investigators propose a single-site, double-blinded, placebo-controlled clinical trial of lavender aromatherapy versus placebo for patient satisfaction in adult women having a surgical abortion before 10 weeks and 0 days gestation. The investigators will evaluate whether lavender aromatherapy is an effective adjunct therapy for patient satisfaction during first trimester surgical abortion. The investigators will measure satisfaction using the Iowa Satisfaction with Anesthesia Scale (ISAS). The investigators hypothesize that women receiving lavender aromatherapy will report higher satisfaction scores compared to women receiving placebo.

Prior studies have investigated the use of aromatherapy in laboring patients, in menstruating women, and in general post-operative populations. No investigations have focused on the use of lavender aromatherapy as an adjunct therapy to paracervical block and/or oral narcotics and anxiolytics in outpatient surgical abortion. This study is novel in investigating patient satisfaction with first trimester surgical abortion using lavender aromatherapy.

The contribution of this proposed research to the literature is significant because current affordable anesthetic adjuncts to opioids and benzodiazepines are limited.

ELIGIBILITY:
Inclusion Criteria:

* Women18 years or older
* Have decide to have a pregnancy termination with no sedation or oral sedation.
* Are less than10 weeks 0 days gestational age with viable pregnancy.
* Agree to being randomized to aromatherapy or placebo

Exclusion Criteria:

* Contraindications or allergies to ibuprofen, lidocaine, or jojoba oil.
* A non-viable intrauterine pregnancy
* A pregnancy greater than or equal to 10 weeks gestational age.
* Adults who are unable to consent or who are currently incarcerated.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Enrollment is limited to patients undergoing a pregnancy termination; therefore, all subjects must be female.
Enrollment: 144 (Actual)
Dates: Start 2021-05-13 (Actual); Primary Completion 2022-04-26 (Actual); Study Completion 2022-04-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leanne Free, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- Comprehensive Women's Health Center, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Free LL, Sheeder J, Cohen RH. Effects of aromatherapy on patient satisfaction with procedural abortion at less than 10 weeks' gestation: A randomized controlled trial. Contraception. 2024 Feb;130:110311. doi: 10.1016/j.contraception.2023.110311. Epub 2023 Oct 17. PMID 37858617
- See also: Guttmacher Institute. "Induced Abortion in the United States," May 3, 2016. — https://www.guttmacher.org/fact-sheet/induced-abortion-united-states
- See also: First-Trimester Surgical Abortion Practices: A Survey of National Abortion Federation Members — https://doi.org/10.1016/j.contraception.2008.11.005
- See also: Micks, Elizabeth A., Alison B. Edelman, Regina Maria Renner, Rongwei Fu, William E. Lambert, Paula H. Bednarek, Mark D. Nichols, Ethan H. Beckley, and Jeffrey T. Jensen. "Hydrocodone-Acetaminophen for Pain Control in First-Trimester Surgical Abortion: — https://doi.org/10.1097/AOG.0b013e31826c32f0
- See also: Ndubisi, Chioma, Antoinette Danvers, Melanie A. Gold, Lisa Morrow, and Carolyn L. Westhoff. "Auricular Acupuncture as an Adjunct for Pain Management during First Trimester Abortion: A Randomized, Double-Blinded, Three Arm Trial." Contraception 99, no. — https://doi.org/10.1016/j.contraception.2018.11.016
- See also: schann, Mary, Jennifer Salcedo, Reni Soon, and Bliss Kaneshiro. "Patient Choice of Adjunctive Nonpharmacologic Pain Management during First-Trimester Abortion: A Randomized Controlled Trial." Contraception 98, no. 3 (September 1, 2018): 205-9. — https://doi.org/10.1016/j.contraception.2018.05.007
- See also: enner, Sallie Stoltz. "Lavandula Angustifolia Miller: English Lavender." Holistic Nursing Practice 23, no. 1 (January 2009): 57-64. — https://journals.lww.com/hnpjournal/abstract/2009/01000/lavandula_angustifolia_miller__english_lavender.9.aspx
- See also: Tanvisut, Rajavadi, Kuntharee Traisrisilp, and Theera Tongsong. "Efficacy of Aromatherapy for Reducing Pain during Labor: A Randomized Controlled Trial." Archives of Gynecology and Obstetrics 297, no. 5 (May 2018): 1145-50 — https://doi.org/10.1007/s00404-018-4700-1
- See also: Upchurch, Dawn M., and Laura Chyu. "Use of Complementary and Alternative Medicine among American Women." Women's Health Issues 15, no. 1 (January 2005): 5-13. — https://doi.org/10.1016/j.whi.2004.08.010
- See also: "Dexter - 2012 - Iowa Satisfaction with Anesthesia Scale.Pdf." Accessed August 24, 2020. — https://www.franklindexter.net/PDF%20Files/IowaSatisfactionAnesthesiaScale.pdf
- See also: Dexter, Franklin. "Iowa Satisfaction with Anesthesia Scale." Korean Journal of Anesthesiology 62, no. 3 (2012): 297. — https://doi.org/10.4097/kjae.2012.62.3.297
- See also: Dexter, Franklin, John Aker, and Will A. Wright. "Development of a Measure of Patient Satisfaction with Monitored Anesthesia Care: The Iowa Satisfaction with Anesthesia Scale." Anesthesiology 87, no. 4 (October 1997): 865-73. — https://doi.org/10.1097/00000542-199710000-00021

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: From May 2021 through April 2022, we assessed 196 participants for eligibility. We excluded 51 potential participants, the majority of whom declined to participate. Of 144 participants consented and enrolled, 73 were randomized to aromatherapy and 71 were randomized to placebo.
Groups:
- Placebo - Jojoba Oil (100% Organic Golden Expeller-pressed Simmondsia Chinensis): Study randomization to lavender aromatherapy or placebo occurred just prior to the initiation of the abortion procedure. A permutated block stratified randomization scheme was utilized so that equal numbers of participants receiving no sedation and PO sedation were randomized to lavender aromatherapy or placebo. 1cc of dilute lavender aromatherapy and placebo will be pre-filled in a 5/8 dram mini amber glass bottle provided to the patient. Immediately prior to procedure start (defined as after receiving antibiotic and emptying bladder), participants were instructed to self-administer the study product. They brought down their personal cloth mask to chin level and rub the study product within the amber glass bottle on their upper lip and nose (left and right ala, alarfacial grooves, and columella). Participants were instructed to take 4 deep breaths and then replace their mask over their nose. The patient then proceeded to the procedure.
  Placebo oil: The placebo group received jojoba oil.
- Investigational Product - A 10% Dilute Lavandula Angustifolia - Jojoba Oil Essential Oil Blend: Study randomization to lavender aromatherapy or placebo occurred just prior to the initiation of the abortion procedure. A permutated block stratified randomization scheme was utilized so that equal numbers of participants receiving no sedation and PO sedation were randomized to lavender aromatherapy or placebo. 1cc of dilute lavender aromatherapy and placebo will be pre-filled in a 5/8 dram mini amber glass bottle provided to the patient. Immediately prior to procedure start (defined as after receiving antibiotic and emptying bladder), participants were instructed to self-administer the study product. They brought down their personal cloth mask to chin level and rub the study product within the amber glass bottle on their upper lip and nose (left and right ala, alarfacial grooves, and columella). Participants were instructed to take 4 deep breaths and then replace their mask over their nose. The patient then proceeded to the procedure.
  Lavender oil: Investigational Product. This group received a 10% lavandula angustafolia diluted in jojoba oil.
Period: Overall Study
Arm/Group | Placebo - Jojoba Oil (100% Organic Golden Expeller-pressed Simmondsia Chinensis) | Investigational Product - A 10% Dilute Lavandula Angustifolia - Jojoba Oil Essential Oil Blend
Started | 71 | 73
Completed | 55 | 57
Not Completed | 16 | 16
Not completed — Physician Decision | 1 | 1
Not completed — Subjects excluded due to enrollment in study prior to registration on ClinicalTrials.gov. | 15 | 15

BASELINE CHARACTERISTICS:
Population: 32 participants were excluded from analysis: 30 were enrolled prior to posting the study on ClinicalTrials.gov; 1 had an undiagnosed ectopic pregnancy, and one had a protocol deviation (did not receive study product).
Groups:
- Total: Total of all reporting groups
Arm/Group | Investigational Product - A 10% Dilute Lavandula Angustifolia - Jojoba Oil Essential Oil Blend | Placebo - Jojoba Oil (100% Organic Golden Expeller-pressed Simmondsia Chinensis) | Total
Number analyzed (Participants) | 57 | 55 | 112
Age, Continuous [Median (Full Range); unit: years] | 27 [18 to 39] | 28 [19 to 40] | 27 [18 to 40]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 55 | 112
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic | 20 | 18 | 38
  Non-Hispanic White | 21 | 22 | 43
  Non-Hispanic Black | 9 | 9 | 18
  Non-Hispanic Other | 7 | 5 | 12
  Prefer not to answer | 0 | 1 | 1
History of [Count of Participants; unit: Participants]
  Vaginal Delivery | 19 | 24 | 43
  Cesarean Delivery | 5 | 7 | 12
  Miscarriage | 13 | 14 | 27
  Medication Abortion | 7 | 3 | 10
  Surgical Abortion | 15 | 18 | 33
  Nulliparous (no SVD or CD) | 33 | 27 | 60
Highest Level of Education [Count of Participants; unit: Participants] — Population: There were 3 non-responders in the aromatherapy group and 1 in the placebo group
  Participants
    Graduated college or graduate school | 24 | 22 | 46
    Less than college (some college, graduated high school, GED, vocational school) | 30 | 32 | 62
    Non-responders | 3 | 1 | 4
Pain with Menses Visual Analog Scale [Median (Full Range); unit: units on a scale] — Baseline menstrual pain was assessed using an unmarked 100mm visual analog scale (VAS) with anchors at 0mm indicating "no pain" and 100mm indicating "severe pain."
  units on a scale | 56 [2 to 99] | 42 [0 to 97] | 51 [0 to 100]
Adjusted State Trait Anxiety Iventory [Median (Full Range); unit: units on a scale] — Additionally, participants completed the State-Trait Anxiety Inventory (STAI) [15], a 40-item self-reported questionnaire to measure current state of anxiety and overall anxiety proneness. All items are rated on a 4-point scale (e.g., from "Almost Never" to "Almost Always") with higher scores indicating greater anxiety. The presence of state or trait anxiety was determined using a cut-off score of 40 which defines a probable clinical diagnosis of anxiety
  units on a scale
    State Anxiety - how a person feels in the moment. Min: 20 max: 80. Higher score is more anxiety . | 43 [24 to 66] | 45 [23 to 68] | 45 [20 to 68]
    Trait Anxiety - how a person generally feels. Min: 20 max: 80. Higher score is more anxiety . | 34 [22 to 65] | 37 [20 to 66] | 36 [20 to 66]

OUTCOME MEASURES:

1. Primary Outcome: Patient Satisfaction With Anesthesia
Description: Difference in patient satisfaction with their abortion experience as measured on the Iowa Satisfaction with Anesthesia Scale (ISAS) following a surgical abortion less than 10 weeks 0 days gestational age between women randomized to lavender aromatherapy versus placebo.
  The self-reported questionnaire consists of 11 items such as "I hurt," "I felt safe," "I had nausea," each assessed on a Likert-type scale ranging from "Disagree very much" to "Agree very much." The responses are then scored from -3 (least satisfied) to +3 (most satisfied) and an average composite score is obtained.
Time Frame: 15 minutes post-procedure
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Investigational Product - A 10% Dilute Lavandula Angustifolia - Jojoba Oil Essential Oil Blend | Placebo - Jojoba Oil (100% Organic Golden Expeller-pressed Simmondsia Chinensis)
Number analyzed (Participants) | 57 | 55
score on a scale | 0.72 (0.96) | 0.46 (0.98)

2. Secondary Outcome: Maximum Procedural Pain
Description: Difference in maximum procedural pain as measured by Visual Analog Scale (VAS) in patients receiving lavender aromatherapy versus placebo. The VAS is presented as a 100-millimeter line with descriptive anchors at each end, "no pain" on the left at 0 centimeters and "pain as bad as it could be" at 100-millimeters. Respondents place a vertical line through the point on the scale that best fits their experience with their procedural pain and that mark is measured as a continuous variable for pain from 0 to 10 (no pain to pain as bad as it could be).
Time Frame: Immediately post-procedure
Population: as for baseline characteristics
Measure: Median (Full Range); unit: millimeters
Arm/Group | Placebo - Jojoba Oil (100% Organic Golden Expeller-pressed Simmondsia Chinensis) | Investigational Product - A 10% Dilute Lavandula Angustifolia - Jojoba Oil Essential Oil Blend
Number analyzed (Participants) | 55 | 57
millimeters | 63 [7 to 97] | 65 [4 to 95]

3. Secondary Outcome: Acceptability
Description: Patient acceptability of lavender aromatherapy as a complementary and alternative medicine used during first trimester surgical abortion as measured through a post-procedure survey.
Time Frame: 11 months
Population: During analysis, participants who "neither agreed or disagreed" were considered not satisfied.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo - Jojoba Oil (100% Organic Golden Expeller-pressed Simmondsia Chinensis) | Investigational Product - A 10% Dilute Lavandula Angustifolia - Jojoba Oil Essential Oil Blend
Number analyzed (Participants) | 55 | 57
Participants
  Agreed inhaling scented was helpful during procedure. | 25 | 41
  Would recommend inhaling scented oil to a friend who needed a procedural abortion. | 31 | 49
  If needed another procedural abortion, would want to inhale scented oil during procedure | 39 | 50

4. Secondary Outcome: Patient Acceptability of Lavender Aromatherapy in Procedural Abortion
Description: We asked: Agreed inhaling scented was helpful during procedure, Would recommend inhaling scented oil to a friend who needed a procedural abortion, If needed another procedural abortion, would want to inhale scented oil during procedure. Participants' acceptability was measured on a 5-point Likert scale (strongly agree, somewhat agree, neither agree or disagree, somewhat disagree, strongly disagree). With strongly agree being a better outcome. Participants who agree with outcome include those who somewhat agree and strongly agree.
Time Frame: 15 minutes post-procedure
Population: During analysis, participants who "neither agreed or disagreed" were considered not satisfied.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo - Jojoba Oil (100% Organic Golden Expeller-pressed Simmondsia Chinensis) | Investigational Product - A 10% Dilute Lavandula Angustifolia - Jojoba Oil Essential Oil Blend
Number analyzed (Participants) | 55 | 57
Participants
  Agreed inhaling scented was helpful during procedure. | 25 | 41
  Would recommend inhaling scented oil to a friend who needed a procedural abortion. | 31 | 49
  If needed another procedural abortion, would want to inhale scented oil during procedure | 39 | 50

ADVERSE EVENTS:
Time Frame: Adverse event data were collect only on the day of the procedure; from time of enrollment into the study until discharge from the clinic.
Description: 32 participants were excluded from analysis: 30 were enrolled prior to posting the study on ClinicalTrials.gov; 1 had an undiagnosed ectopic pregnancy, and one had a protocol deviation (did not receive study product).
Arm/Group | Placebo - Jojoba Oil (100% Organic Golden Expeller-pressed Simmondsia Chinensis) | Investigational Product - A 10% Dilute Lavandula Angustifolia - Jojoba Oil Essential Oil Blend
All-Cause Mortality (participants affected / at risk) | 0/71 | 0/73
Serious Adverse Events (participants affected / at risk) | 0/71 | 0/73
Other Adverse Events (participants affected / at risk) | 0/71 | 0/73

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-10-26): https://cdn.clinicaltrials.gov/large-docs/00/NCT04969900/Prot_SAP_000.pdf